CLINICAL TRIAL: NCT02911545
Title: Non-vitamin K Oral Anticoagulants in Cardioversion of Atrial Fibrillation. FinCV3
Brief Title: Non-vitamin K Oral Anticoagulants in Cardioversion
Acronym: FinCV3
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Turku (Other)
Responsible Party: Principal Investigator, Mika Lehto, MD, PhD, cardiologist, Helsinki University Central Hospital
Other Study IDs: FinCV3
Record Dates: First submitted 2016-09-16; First posted 2016-09-22 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Anticoagulation; Cardioversion
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Non-vitamin K oral anticoagulants (NOAC) have been shown to be safe and effective alternatives to warfarin for stroke prevention in patients with nonvalvular AF (NVAF). There are yet limited real life data on outcomes following elective cardioversion in AF patients treated with NOACs. The aim of this study is to investigate the complications and the use of NOACs in AF patients undergoing cardioversion.

ELIGIBILITY:
Inclusion Criteria:

* AF patients undergoing cardioversion

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: AF patients undergoing cardioversion.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2011-10; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Incidence and predictors of thromboembolic complications | 31 days after cardioversion of persistent AF
Incidence and predictors of bleeding | 31 days after cardioversion of persistent AF

SECONDARY OUTCOMES:
Number of recurrence of AF | 31 days after cardioversion of persistent AF
Hemodynamic complications of cardioversion | 31 days after cardioversion of persistent AF

CONTACTS AND LOCATIONS:
Overall Officials: Mika Lehto, MD, PhD, Principal Investigator — Helsinki University Central Hospital

IPD SHARING:
Plan to Share IPD: No